CLINICAL TRIAL: NCT01562860
Title: The Influence of Pronator Teres Release in the Treatment of Median Nerve Compression Neuropathy: A Randomized Prospective Study
Brief Title: Influence of Pronator Teres Release on Treatment of Median Nerve Compression Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.0039
Record Dates: First submitted 2011-08-08; First posted 2012-03-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Median Nerve Compression
Keywords: median nerve; carpal tunnel syndrome; Pronator Teres Release
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carpal Tunnel and Pronator Teres Release (Active Comparator): Patients enrolled in this arm of the study will have both surgical procedures performed at the same time
  Interventions: Procedure: dual compression release
- Carpal Tunnel Release only (Active Comparator): Patients enrolled in this arm will have only Carpal Tunnel Release performed. In they still have symptoms of median nerve neuropathy, they will be scheduled for an additional procedure to release the pronator Teres in a separate surgery.
  Interventions: Procedure: Pronator Teres Release; Procedure: dual compression release; Procedure: median nerve release only

INTERVENTIONS:
Procedure: Pronator Teres Release — Surgical release of median nerve compression
  Other Names: carpal tunnel release
  Arms: Carpal Tunnel Release only
Procedure: dual compression release — Both the carpal tunnel compression and the pronator teres compression will be released on the same day.
  Arms: Carpal Tunnel Release only
Procedure: dual compression release — both procedures will be done on the same day
  Arms: Carpal Tunnel and Pronator Teres Release
Procedure: median nerve release only — only the carpal tunnel compression is released
  Arms: Carpal Tunnel Release only

SUMMARY:
The investigators are comparing two standard of care procedures which can be performed at the same time, or sequentially. The hypothesis being tested is whether simultaneous release of both the carpal Tunnel and the Pronator Teres results in a better outcome in terms of symptom relief and recurrence than Carpal Tunnel Release alone when signs and symptoms of both carpal tunnel and pronator Teres syndromes are present.

ELIGIBILITY:
* Inclusion Criteria: Positive Tinnels signs over the median nerve at the Carpal Tunnel and Pronator Teres
* Normal two point discrimination
* Over the age of 18 and under the age of 65

Exclusion Criteria:

* Peripheral neuropathy of the median nerve secondary to trauma
* Presence of thoracic outlet syndrome
* Presence of cervical disk disease
* Under the age of 18 and over the age of 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Symptom severity and functional status score (Brigham and Women's Carpal Tunnel Questionnaire) | 12 months
  The primary outcome measure will be the difference between the pre and post operative assessments of the questionnaire, which will represent the degree of improvement as result of the surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Ozyurekoglu, MD, Principal Investigator — Christine M. Kleinert Institute for Hand and Microsurgery
Locations (1):
- Christine M. Kleinert Institute for Hand and Microsurgery, Louisville, Kentucky, United States